CLINICAL TRIAL: NCT07241234
Title: A Phase 1b, Open-label, Multicenter, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of AG-181 in Subjects With Phenylketonuria
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AG-181 in Subjects With Phenylketonuria
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AG181-C-002; 2025-522630-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: AG-181 (Experimental): Subjects will receive AG-181 from Day 1 to Day 28.
  Interventions: Drug: AG-181
- Cohort 2 (Optional Cohort): AG-181 (Experimental): Subjects will receive AG-181.
  Interventions: Drug: AG-181

INTERVENTIONS:
Drug: AG-181 — AG-181 film-coated tablets

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AG-181 in subjects with Phenylketonuria (PKU).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PKU, defined as documented presence of 2 mutant alleles in the phenylalanine hydroxylase (PAH) gene, of which at least 1 is the R408W mutation, as determined during Screening per the genotyping performed by the study central genotyping laboratory.
* At least 1 plasma Phe concentration greater than (>) 600 micromoles per liter (μmol/L) in the 52 weeks before providing informed consent.
* Average concentration of plasma Phe > 600 μmol/L in Phe samples taken during Screening, with no individual assessment below 360 μmol/L. Any Phe samples taken after Day -20 will not be included.
* Body mass index (BMI) greater than or equal to (≥) 18.0 kilograms per meter square (kg/m^2) to lesser than or equal to (≤) 35.0 kg/m^2 and weight ≥ 50 kilograms (kg) at any time during the Screening Period.
* Documented approval from a dietitian confirming that the subject can maintain their diet consistent in protein and Phe intake throughout the study as outlined in the Diet Manual.

Key Exclusion Criteria:

* Prior exposure to AG-181.
* Receiving inhibitors of P-glycoprotein (P-gp) that have not been stopped for ≥ 5 days or a timeframe equivalent to 5 half-lives (whichever is longer) before administration of the first dose of study drug.
* Receiving products that are strong inhibitors or strong inducers of cytochrome P450 CYP1A2, CYP2C8, or CYP3A that have not been stopped for ≥ 28 days before administration of the first dose of study drug.
* Receiving treatment with an acid-reducing agent, including but not limited to proton pump inhibitors and H2 blockers. Short-acting acid-reducing agents such as calcium carbonate are permitted.
* Any preexisting condition that could (in the opinion of the Investigator) interfere with gastrointestinal anatomy or motility that may disrupt the absorption, metabolism, and/or excretion of the study drug.
* Any preexisting condition that could (in the opinion of the Investigator) interfere with hepatic or renal function that may disrupt the absorption, metabolism, and/or excretion of the study drug.
* Inability to tolerate oral medication.
* Unwillingness to washout from tetrahydrobiopterin (BH4) supplementation (eg, sapropterin dihydrochloride, Kuvan), pegvaliase-pqpz (Palynziq), or any other PKU therapy by Day -30 during Screening.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01-17 (Estimated); Study Completion 2028-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events (AEs) and Serious Adverse Events (SAEs) by Type, Severity, and Relationship to the Study Drug | Up to Day 42

SECONDARY OUTCOMES:
Plasma Concentration of AG-181 | Up to Day 28
Maximum Concentration (Cmax) of AG-181 | Up to Day 28
Time to Maximum (Peak) Concentration (Tmax) of AG-181 | Up to Day 28
Area Under the Concentration-Time Curve (AUC) of AG-181 | Up to Day 28
Apparent Total Body Clearance (CL/F) of AG-181 | Up to Day 28
Apparent Volume of Distribution in the Terminal Phase (Vz/F) of AG-181 | Up to Day 28
Change From Baseline in Phenylalanine (Phe) Concentration | Baseline up to Day 28

IPD SHARING:
Plan to Share IPD: No